CLINICAL TRIAL: NCT06366373
Title: Reducing Stigma Through a Mental Health Art Exhibition and Its Printed Brochure: an Social-contact Intervention Study
Brief Title: Reducing Stigma Through a Mental Health Art Exhibition and Its Printed Brochure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan University (Other)
Collaborators: Central South University (Other); Qixi Charity (Unknown)
Responsible Party: Principal Investigator, Wei Zhou, Associate Professor, Hunan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 531118232022
Record Dates: First submitted 2024-03-30; First posted 2024-04-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Issue
Keywords: mental health; stigma; discrimination; social contact
MeSH Terms: conditions — Psychological Well-Being; Social Stigma

STUDY DESIGN:
Intervention Model Description: The interventional study model for this clinical trial is a two-phase experimental design.
  At Phase One, a single-arm pre-post study design will be adopted. Specifically, the intervention is the exhibition, organized by "Qixi Charity," will publicly display offline artworks reflecting the diverse dimensions of mental health and ill-health.
  At Phase Two, a multiple-arm pre-post study design will be adopted. Specifically, the intervention become the printed brochure of the exhibition and its effect will be compared with a traditional health education brochure and a postcard as a placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- an exhibition group (Experimental): At Phase One, participants of this group are those who attend the offline art exhibition. At Phase Two, participants of this group are those who cannot attend the offline exhibition and will be provied with a printed brochure of the exhibition.
  Interventions: Other: A mental health art exhibition
- an education group (Active Comparator): At Phase Two, participants in this group are those who are unable to attend the offline art exhibition but will be provided with printed/online education materials
  Interventions: Other: printed or online education materials
- Control Group (No Intervention): At Phase Two, participants in this group are those who cannot attend the exhibition offline and will be provided with a postcard.

INTERVENTIONS:
Other: A mental health art exhibition — The specific intervention measure is the Second Mental Health Art Science Exhibition scheduled to take place in Wuhan, China from April 27 to May 27, 2024. Organized by "Qixi Charity", an NGO led by individuals with lived experience of mental disorders, as well as their family members and friends, the exhibition will feature offline artworks created by these individuals and other contributors. The exhibited artworks aim to reflect the diverse dimensions of mental health and ill-health.
  Arms: an exhibition group
Other: printed or online education materials — The specific intervention measure is to provide printed or online education materials within the first month after the baseline survey
  Arms: an education group

SUMMARY:
Mental health art exhibitions, as an intervention strategy integrating artistic expression and social contact, have the potential to positively impact the elimination of stigma and discrimination associated with mental health problems. Based on a two-phase experimental design, this study aims to evaluate the effect of a real-world mental health art exhibition (Phase One) and its printed brochure (Phase Two) on stigma/discrimination and related outcomes, such as mental health literacy. The evaluation will encompass three categories of people: those with lived experience of mental disorders, family members and friends of those with lived experience, and the general public. Qualitative methods, such as in-depth interviews, will also be used for the evaluation.

DETAILED DESCRIPTION:
Mental health art exhibitions, as an intervention strategy integrating artistic expression and social contact, have the potential to positively impact the elimination of stigma and discrimination associated with mental health problems. Based on a two-phase experimental design, this study aims to evaluate the effect of a real-world mental health art exhibition (Phase One) and its printed brochure (Phase Two) on stigma/discrimination and related outcomes, such as mental health literacy. The evaluation will encompass three categories of people: those with lived experience of mental disorders, family members and friends of those with lived experience, and the general public. Qualitative methods, such as in-depth interviews, will also be used for the evaluation.

The intervention measure is the Second Mental Health Art Science Exhibition scheduled to take place in Wuhan, China from April 27 to May 14, 2024. Organized by "Qixi Charity", an NGO led by individuals with lived experience of mental disorders, as well as their family members and friends, the exhibition will feature offline artworks created by these individuals and other contributors. The exhibited artworks aim to reflect the diverse dimensions of mental health and ill-health.

At Phase One, the effect of the real-world exhibition is evaluated through a single-arm pre-post study design. The adult audience, who are individuals with lived experience of mental disorders, or family members and friends of those with lived experience, or the general public, will be recruited as the experimental group, and they will be surveyed three times: (1) a baseline survey before the interventions (T0); (2) a follow-up survey in the first month after the interventions (T1); (3) a follow-up survey in the sixth month after the interventions (T2). Additionally, the study will perform text analysis of media reports and social media discussions related to the exhibition to supplement the assessment of its social impact.

Due to the high costs and limited feasibility of widespread implementation of the real-world Mental Health Art Exhibition, the intervention was then adapted to a printed exhibition brochure. At Phase Two, the effect of the brochure intervention in reducing stigma and other related outcomes will be assessed and compared with a traditional health education brochure and a postcard as a placebo. Individuals with lived experience of mental disorders, or family members and friends of those with lived experience, or the general public, who do not visit the exhibition of Phase One, will be recurited. After that, individuals with lived experience of mental disorders and their family members or friends will be cluster-randomized to either the exhibition brochure group or the control group (the latter typically receives or seeks out traditional health education materials during healthcare visits). As for the general public will be cluster-randomized into three groups: (1) the exhibition brochure group, (2) the traditional health education brochure group, and (3) the control group. Effectiveness will be evaluated through three surveys: (1) a baseline survey before the interventions (T0); (2) a follow-up survey one month after the interventions (T1); and (3) a follow-up survey six months after the interventions (T2).

ELIGIBILITY:
General Inclusion Criteria:

* Adults aged 18 and above

General Exclusion Criteria:

* Individuals who are unable to understand the content of the questionnaire due to illness and other factors
* Mental health professionals, including psychiatrists, psychologists, nurses, social workers and medical students

Additional Inclusion Criteria for Phase One:

* Individuals who attend the exhibition offline

Additional Inclusion Criteria for Phase Two:

* Individuals who did not visit the exhibition of Phase One

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Stigma/discrimination regarding mental disorders | Time point 0: before the exhibition; Time point 1: within the first month after the exhibition; Time point 2: the sixth month after the exhibition
  Individuals with lived experience of mental disorders: internalized stigma of mental illness scale (ISMI-29), the perceived devaluation discrimination scale (PDD-12) Family members and friends of those with lived experience: affiliate stigma scale (ASS-22), the perceived devaluation discrimination scale (PDD-12) The general public: community attitudes toward mental ill scale (CAMI-20), attribution questionnaire (AQ-9), the perceived devaluation discrimination scale (PDD-12)

SECONDARY OUTCOMES:
mental health literacy | Time point 0: before the exhibition; Time point 1: within the first month after the exhibition; Time point 2: the sixth month after the exhibition
  All participants: mental health and care knowledge questionnaire (MHCK-16)

OTHER OUTCOMES:
Willingness to pay | T2: six months after the interventions (T2)
  Individuals with lived experience of mental disorders & family members and friends of those with lived experience: maximum and minimum amount of money willing to pay for treating the suffering mental health conditions The general public: maximum and minimum amount of money willing to pay for treating 2 mental health conditions and 2 general health conditions in vignettes

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhou, Ph.D., Principal Investigator — Hunan University
Locations (3):
- China (3):
  - Qixi Charity, Wuhan, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No